CLINICAL TRIAL: NCT00734552
Title: Randomized, Open-Label, Prospective Study to Evaluate the Protective Effect of α-Keto Acid With Low-protein Diet on Residual Renal Function (RRF) in Peritoneal Dialysis Patients
Brief Title: Study to Evaluate the Protective Effect of α-Keto Acid With Low-protein Diet on Renal Function in PD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xue Qing Yu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSU-KAPDRRF
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Peritoneal Dialysis
Keywords: Continuous Ambulatory Peritoneal Dialysis; α-Keto Acid; Low Protein Diet; Residual Renal Function
MeSH Terms: interventions — Diet, Protein-Restricted; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): α-Keto Acid plus low protein diet
  Interventions: Dietary Supplement: α-Keto Acid with low protein diet
- 2 (Other): Normal protein diet
  Interventions: Dietary Supplement: Normal protein diet

INTERVENTIONS:
Dietary Supplement: α-Keto Acid with low protein diet — Compound α-Keto Acid: The daily dose of compound α-Keto Acid is 0.1/kg/d. The total daily dose will be divided into three times a day.
  Low Protein Diet: Diet contain protein 0.8g/kg/d.
  Other Names: Test Group
  Arms: 1
Dietary Supplement: Normal protein diet — Diet contain protein 1.0-1.2 g/kg/d.
  Other Names: Control Group
  Arms: 2

SUMMARY:
This randomized, open-label, prospective study will evaluate the renal effective effect of compound α-Keto Acid plus low protein diet in PD Patients.

DETAILED DESCRIPTION:
Residual renal function (RRF) is associated with cardiovascular complication, nutritional status, incidence of peritonitis, and quality of life in peritoneal dialysis (PD) patients. Therefore, RRF is an important determinant of mortality and morbidity in PD patients.

Previous studies have suggested that dietary protein restriction supplemented with compound keto/amino acids may slow the loss of RRF in chronic kidney disease patients. However, there is very few reports to address the effect of compound keto/amino acid supplementation in RRF in PD patients.

The aim of this study is to evaluate the protective effect of compound α-Keto Acid plus low protein diet in RRF in PD Patients.This is a randomized, open-label, prospective study. 100 patients who meet Inclusion/Exclusion criteria will be randomized into α-Keto Acid group or control group at the ratio of 1:1. α-Keto Acid group will use compound α-Keto Acid plus low protein diet, while control group will use normal protein diet.Compound α-Keto Acid dosage is 0.1/kg/d daily. The effect of compound α-Keto Acid plus low protein diet in RRF will be evaluated after 1 year treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients on PD at least one month prior to study entry.
2. Subjects of either sex, more than 20 years old, the range of age is 20 to 75 year old.
3. Residual GFR ≥3 ml/min/1.73m2.
4. Residual urine volume ≥ 500 ml/24h.
5. No history of taking α-Keto Acid within 2 weeks.
6. Subjects who agree to participate in the study and sign the informed consent.

Exclusion Criteria:

1. History of peritonitis or other infection within one month.
2. History of taking drug which may affect amino acid metabolism within one month.
3. Incapable of following study requirements to control diet.
4. With severe cardiovascular disease, chronic liver disease, dyscrasia, psychiatric disorder, alcohol or drug abuse.
5. Participation in another clinic trial within one month prior to screening.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
The longitudinal change in residual glomerular filtration rate (GFR),residual urine volume | Every 3 months

SECONDARY OUTCOMES:
Peritoneal membrane transport characteristics,cardiovascular events,nutritional status,hospitalization, peritonitis episodes, any adverse drug effects. | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Xueqing Yu, M.D. & Ph.D., Principal Investigator — 1st Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The 1st Affiliated Hospital, Sun Yet-sen University, Guangzhou, Guangdong, China